CLINICAL TRIAL: NCT02645370
Title: Efficacy and Safety of Danzhen in the Preventive Treatment of Migraine:A Prospective "Real-World" Study.
Brief Title: Efficacy and Safety of Danzhen
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Ecion Pharmaceutical CO..LTD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Xijing-APP-CER
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Migraine
Keywords: Migraine; Danzhen; Topiramate; Headache diary APP; preventive treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator:Topiramate (Active Comparator): The treatment with TPM is initiated at a 50 mg daily dose and sequentially increase every 7 days, as tolerated, in 25 mg increments up to a target dose of 150 mg total/day.
  Interventions: Drug: Topiramate
- Experimental:Danzhen (Experimental): The treatment with Danzhen is 3 tablets triple daily.
  Interventions: Drug: Danzhen

INTERVENTIONS:
Drug: Danzhen
  Arms: Experimental:Danzhen
Drug: Topiramate
  Other Names: TPM
  Arms: Active Comparator:Topiramate

SUMMARY:
The purpose is to evaluate the effectiveness and safety profile of Danzhen for the prophylaxis of migraine in a "real-world" setting.

DETAILED DESCRIPTION:
In adults between 18- and 65-years in China,the prevalence of migraine is 9.3% in general. Migraine is a heterogeneous condition that may produce a range of symptom profiles and various degrees of disability.The disability resulting from migraine can be severe imposing a considerable health burden upon the sufferer and society. The purpose of this study, using topiramate as the control, is to evaluate the effectiveness and safety of Danzhen for the prophylaxis of migraine in a "real-world"setting.Patients are asked to maintain a detailed headache diary via headache diary APP throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than or equal to 18 years and less than 70 years.
* The diagnosis of migraine is made according to 2004 The International Classification of Headache Disorders: 2nd edition (ICHD-II) .
* Consent form signed by the participant or his/her authorized surrogate.

Exclusion Criteria:

* Patients had primary or secondary headache disorders other than migraine.
* Female subjects of childbearing age will be excluded if they were pregnant, lactating or planning apregnancy in the next year or if they were not using an adequate form of birth control.
* Patients will be excluded if they had significant medical or psychiatric disease,or taking another antidepressant for any reason and not able to discontinue.
* Patients used other preventive pharmacological agents during the 1 month prior to baseline period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
A 50% or greater reduction in headache days/month during the third treatment month of maintenance phase relative to baseline phase with one of the study drugs. | at baseline phase/the third treatment month of maintenance phase

SECONDARY OUTCOMES:
The decrease of disability days of migraine/month | at baseline phase/the third treatment month of maintenance phase
The decrease of numbers of rescue medication doses used/month | at baseline phase/the third treatment month of maintenance phase
A 30% or greater reduction in headache time | at baseline phase/the third treatment month of maintenance phase
The percentage of discontinued the drug because of side effects | at the third treatment month of maintenance phase
Beck Depression Inventory (BDI) scores | at the third treatment month of maintenance phase
Compliance | at the third treatment month of maintenance phase

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China